CLINICAL TRIAL: NCT00370851
Title: Intravitreal Bevasizumab VS Sham Treatment in Acute BRVO: A Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8532
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Retinal Disease
Keywords: intravitreal Avastin; BRVO; Macular edema
MeSH Terms: conditions — Retinal Diseases; Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Intravitreal injection of Avastin
  Interventions: Drug: Avastin (Bevacizumab)
- 2 (Sham Comparator)
  Interventions: Drug: Avastin (Bevacizumab)

INTERVENTIONS:
Drug: Avastin (Bevacizumab) — Intravitreal injection of 125 mg Avastin

SUMMARY:
In this study we intend to evaluate the outcome of intravitreal avastin on improving the visual acuity and macular edema and late complications of BRVO like NVD and NVE

DETAILED DESCRIPTION:
After diabetic retinopathy, vein occlusion is the second most common retinovascular disease. According to BVO study the only effective management of it is macular photocoagulation for macular thickening that persist after 3 months.But we may miss a golden time which resulted to photoreceptor degeneration due to macular edema during this period. VEGF inhibitors newly have been shown that may be effective on a wide range of retinovascular diseases that resulted to macular edema or new vessels formation. In this study we aim to show the outcomes of one of this VEGF inhibitors (bevacizumab) on complications of BRVO in a sham controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute BRVO with less than three month duration

Exclusion Criteria:

* vision less than 20/320 and vison more than 20/50
* duration more than 3 months
* history of glaucoma and diabetic retinopathy
* any media opacity that prevent funduscopy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | At 12 week
Macular thickness by OCT | At 12 week

SECONDARY OUTCOMES:
Need for macular photocuagulation | At 12th week
Incidence of new vessel formation | At 12th week

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Moradian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Siamak Moradian, MD, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Moradian S, Faghihi H, Sadeghi B, Piri N, Ahmadieh H, Soheilian M, Dehghan MH, Azarmina M, Esfahani MR. Intravitreal bevacizumab vs. sham treatment in acute branch retinal vein occlusion with macular edema: results at 3 months (Report 1). Graefes Arch Clin Exp Ophthalmol. 2011 Feb;249(2):193-200. doi: 10.1007/s00417-010-1440-8. Epub 2010 Aug 18. PMID 21337043